CLINICAL TRIAL: NCT02657759
Title: EFFECTS OF CARDICHOL, AN HERBAL DIETARY SUPPLEMENT, IN MODERATE HYPERCHOLESTEROLEMIA
Acronym: CARDICHOL 1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Direct Plantes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DPlantes
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: HYPERCHOLESTEROLEMIA
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CARDICHOL (Experimental): Food supplement formula in shape of pill called CARDICHOL. 2 pills daily during 12 weeks (from visit V1 to visit V4). One pill immediately before, after or during breakfast and lunch.
  Interventions: Dietary Supplement: CARDICHOL
- Placebo (Placebo Comparator): placebo with the same characteristics, appearance, packaging, and composition as the active formula, except for active ingredients replaced by dicalcium phosphate and flavouring substances.
  2 pills daily during 12 weeks (from visit V1 to visit V4). One pill immediately before, after or during breakfast and lunch.
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: CARDICHOL
  Arms: CARDICHOL
Dietary Supplement: PLACEBO
  Arms: Placebo

SUMMARY:
This research aims to evaluate the effect of CARDICHOL chronic consumption (12 weeks) on lipid metabolism and especially on blood LDL cholesterol in volunteers with moderate hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to the study, male and female volunteers will have to fulfill the following criteria (assessment based on the medical examination performed at V0 with a checking at V1):

* Age between 18 and 65 years (limits included).
* BMI between 18,5 and 30 kg/m² (limits excluded).
* For women: Non menopausal with the same reliable contraception since at least three cycles before the beginning of the study and agreeing to keep it during the entire duration of the study (condom alone without spermicide gel excluded) or menopausal without or with hormone replacement therapy (oestrogenic replacement therapy begun from less than 3 month excluded).
* Good general and mental health with in the opinion of the investigator: no clinically significant and relevant abnormalities of medical history or physical examination.
* Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form.
* Affiliated with a social security scheme.
* Agree to be registered on the volunteers in biomedical research file.

After V0 biological analysis the subjects will be eligible to the study on the following criteria:

- Fasting blood LDLc level (Friedewald estimation method) between 1,3 and 2,2g/L (limits included with ± 2% tolerated around).

A re-screening can occur from 2 months after the exit of study for failure to comply with the one or more of the eligibility criteria listed above.

Exclusion Criteria:

Volunteers with the following criteria will be considered as non eligible to the study (assessment based on the medical examination performed at V0 with a checking at V1):

* Suffering from a metabolic disorder such as diabetes, uncontrolled thyroidal trouble or other metabolic disorder.
* Suffering from a severe chronic disease (e.g. cancer, HIV, renal failure, hepatic or biliary disorders ongoing, chronic inflammatory digestive disease, arthritis or other chronic respiratory trouble, etc.) or gastrointestinal disorders found to be inconsistent with the conduct of the study by the investigator (e.g. celiac disease).
* With a history of ischemic cardiovascular event or, during the previous 6 months a surgical procedure.
* Suffering from an uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg).
* With a known or suspected food allergy or intolerance or hypersensitivity to any of the study products' ingredient.
* Pregnant or lactating women or intending to become pregnant within 4 months ahead.
* Requiring a cholesterol lowering by immediate pharmacologic intervention according to the current recommendations (AFSSAPS 2005).
* Under lipid-lowering treatment (e.g. statins, fibrates, ezetimibe, bile acid sequestrants, niacin, etc.) or stopped less than 4 months before the randomization.
* Under medication which could affect blood lipid parameters (e.g. long-term corticosteroid systemic drug, systemic antibodies, androgens or phenytoin, etc.) or stopped less than 1 month before the randomization (stable long-term treatment with beta blocker or thiazide diuretics tolerated).
* Regular intake of dietary supplements or "health foods" which are known to decrease LDLc or triglycerides (e.g. rich in plant stanol or sterol like PRO-ACTIV or DANACOL products, red yeast rice, policosanol, capsules containing omega-3 fatty acids from fish oils, etc.) or stopped less than 3 months before the randomization.
* Under treatment or dietary supplement which could significantly affect parameter(s) followed during the study according to the investigator or stopped in a too short period before the randomization.
* With significant change in food habits or in physical activity in the 3 months before randomization or not agreeing to keep them unchanged throughout the study.
* With reported body weight variation > 5% in the 3 months prior the randomization or with a hyper or hypocaloric diet planned in the next 4 months.
* With a personal history of anorexia nervosa, bulimia or significant eating disorders according to the investigator.
* Consuming more than 3 standard drinks of alcoholic beverage for men or 2 standard drinks daily for women or not agreeing to keep his alcohol consumption habits unchanged throughout the study.
* Smoking more than 10 cigarettes daily or not agreeing to keep his smoking habits unchanged throughout the study.
* Having a lifestyle deemed incompatible with the study according to the investigator including high level physical activity (defined as more than 10 hours of significant physical activity a week, walking excluded).
* Who made a blood donation in the 3 months before the randomization or intending to make it within 5 months ahead.
* Taking part in another clinical trial or being in the exclusion period of a previous clinical trial.
* Having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros.
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision.
* Presenting a psychological or linguistic incapability to sign the informed consent.
* Impossible to contact in case of emergency.

After V0 biological analysis the subjects will be considered as non eligible to the study on the following criteria:

* Fasting blood glucose level > 1,26 g/L (6,99 mmol/L).
* Fasting blood triglycerides > 3,5 g/L (3,95 mmol/L).
* Fasting blood TC > 4,5 g/L or HDLc < 0,1 g/L with an abnormality judged as clinically significant according to the investigator.
* Blood AST > 1,68 µkat/L, ALT > 1,70 µkat/L or GGT > 2,55 µkat/L (values corresponding to 2,5xULN).
* Blood urea > 12,11 mmol/L (value corresponding to 1,5xULN) or creatinine > 125 µmol/L.
* Complete blood count with hemoglobin < 11 g/L or leucocytes < 3000 / mm3 or leucocytes > 16000 /mm3 or clinically significant abnormality according to the investigator.

A re-screening can occur from 2 months after the exit of study for failure to comply with the one or more of the eligibility criteria listed above.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Change of the fasting blood LDL cholesterol NCEP concentration | 8 weeks

SECONDARY OUTCOMES:
Change of the fasting blood LDL cholesterol concentration (NCEP and Friedewald estimation methods) | 4 weeks
Change of the fasting blood LDL cholesterol concentration (Friedewald estimation method) | 8 weeks
Change of the fasting blood LDL cholesterol concentration (NCEP and Friedewald estimation methods) | 12 weeks
Change of the fasting blood HDL cholesterol concentration (NCEP and direct methods) | 4 weeks
Change of the fasting blood HDL cholesterol concentration (NCEP and direct methods) | 8 weeks
Change of the fasting blood HDL cholesterol concentration (NCEP and direct methods) | 12 weeks
Change of the fasting blood total cholesterol concentration | 4 weeks
Change of the fasting blood total cholesterol concentration | 8 weeks
Change of the fasting blood total cholesterol concentration | 12 weeks
Change of the fasting blood triglycerides concentration | 4 weeks
Change of the fasting blood triglycerides concentration | 8 weeks
Change of the fasting blood tiglycerides concentration | 12 weeks
Change of the fasting blood apolipoprotein B100 concentration | 4 weeks
Change of the fasting blood apolipoprotein B100 concentration | 8 weeks
Change of the fasting blood apolipoprotein B100 concentration | 12 weeks
Change of the fasting blood glucose concentration | 4 weeks
Change of the fasting blood glucose concentration | 8 weeks
Change of the fasting blood glucose concentration | 12 weeks
Change of the fasting blood hsCRP concentration | 4 weeks
Change of the fasting blood hsCRP concentration | 8 weeks
Change of the fasting blood hsCRP concentration | 12 weeks
Change of the ratio of fasting blood concentrations LDLox/LDLc (NCEP method) | 8 weeks
Change of the fasting arylesterase activity (PON-1) in blood | 8 weeks

OTHER OUTCOMES:
Complete blood count | 12 weeks
Blood Aspartate Amino Transferase | 12 weeks
Blood Alanine Amino Transferase | 12 weeks
Blood Gamma Glutamyl Transpeptidase | 12 weeks
Blood total bilirubin | 12 weeks
Blood creatinine | 12 weeks
Blood urea | 12 weeks
Blood Lactate Deshydrogenase | 12 weeks
Blood Creatine Kinase | 12 weeks
Glycated hemoglobin | 12 weeks
Heart rate | 12 weeks
Systolic Blood Pressure | 12 weeks
Diastolic Blood Pressure | 12 weeks
Body weight | 4 weeks
Body weight | 8 weeks
Body weight | 12 weeks
Physical Activity Score | 4 weeks
Physical Activity Score | 8 weeks
Physical Activity Score | 12 weeks
Total energy intake | 8 weeks
Percentage of energy intake from fat | 8 weeks
Dietary fiber intake | 8 weeks
Saturated Fatty Acids intake | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrice CHAUVEAU, Study Director — BioFortis
Locations (1):
- Biofortis, Saint-Herblain, France

IPD SHARING:
Plan to Share IPD: Undecided